CLINICAL TRIAL: NCT01795092
Title: A Randomized-controlled Study to Assess the Impact of Dermatology Consultations on Reducing Admissions for Patients Presenting to Internal Medicine Clinics for Possible Cellulitis
Brief Title: A Study Assessing the Impact of Dermatology Consultation in Patients Presenting With Possible Cellulitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniela Kroshinsky, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008A058574; 2008A058574 (Other Grant/Funding Number: Dermatology Foundation)
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Cellulitis
Keywords: Cellulitis; Outpatient Medicine
MeSH Terms: conditions — Cellulitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Those in the control group do not obtain a dermatology evaluation and will be assessed and treated by their primary care provider. We will perform a chart review two weeks after presentation to assess for admission versus discharge home from clinic and outcome.
- Dermatology consultation (Experimental): Patients randomized to the treatment group will obtain a dermatology evaluation at the primary care physician's office and will be sent to the Emergency Department (ED) or discharged home with outpatient dermatology follow-up in 2-3 days to assess their condition. Patients who are evaluated by a dermatologist and require hospitalization will have their transition to the ED managed by the dermatologist. Patients who are admitted after the initial outpatient discharge or at the follow-up visit will be considered treatment failures. A medical record review will be performed for patients in the treatment group two weeks after initial evaluation at the internal medicine clinic.
  Interventions: Other: Dermatology Consultation

INTERVENTIONS:
Other: Dermatology Consultation — A dermatology consultation will be conducted on patients randomized to this group.
  Arms: Dermatology consultation

SUMMARY:
This is a randomized, controlled study to compare patients evaluated by primary care physicians alone versus patients who are additionally evaluated by a dermatologist at the primary care physician"s office, aiming to demonstrate that visits to the primary care physician"s (PCP) office that involve both the PCP and an on-site dermatology consultation will reduce hospital admission rates. The hypothesis of this study is that obtaining outpatient dermatology consultations during a patient"s initial presentation to a primary care office will reduce admissions for cellulitis with accuracy. The primary objective will be to measure the difference in the proportion of patients requiring hospital admission utilizing a dermatology consultation at the PCP"s office (active arm) versus primary care evaluation alone (control arm) by calculating risk ratios and risk differences. The risk of admission for each arm will be assessed once the study has been completed. The secondary endpoint will be admission versus discharge home at a dermatology follow-up visit to assess accuracy of initial assessment. An additional endpoint will be to determine if any differences in frequencies of cellulitis and admission exist based on age and immunosuppression. Exploratory analyses will assess the percentage of patients with a concomitant known predisposing factor for recurrent cellulitis such as lymphedema, leg ulceration, tinea pedis, or onychomycosis, as well as the association of fever >100.5 F and a history of a prior episode of cellulitis.

DETAILED DESCRIPTION:
Patients to be enrolled in the study will be those that present to outpatient internal medicine clinic and are identified by primary care physicians as having pain, redness, and swelling of the skin that the physician believes may represent cellulitis. Patient recruitment will occur at five Massachusetts General Hospital (MGH) outpatient internal medicine clinical sites: Medical Walk-In, Internal Medicine Associates, Bulfinch Medical Group, Senior Health, and Women's health. Patients with abnormal vital signs will be excluded, specifically systolic blood pressure <90 mmHg, diastolic blood pressure <80 mmHg, heart rate greater than 90 beats per minute or less than 50 beats per minute, respiratory rate greater than 20, or temperature >100.5 F. In addition, any patients with a history of transplantation must be more than six months after initial transplant with no treated episodes of acute rejection in the last 90 days, no use of antithymocyte globulin or campath to treat rejection in the last 6 months, or more than 20 mg/day of prednisone for more than 30 days.

Once a patient is identified with potential cellulitis who is a candidate for outpatient treatment, the primary care physician will then approach them regarding their interest in entering our study. Patients will be randomized during this initial presentation to their primary care physician. The patients randomized to the treatment group will obtain a dermatology evaluation at the primary care physician"s office and will be sent to the Emergency Department or discharged home with outpatient dermatology follow-up in two to three days to assess for improvement in their condition versus no change or worsening that requires transfer to the Emergency Department. Patients who are evaluated by a dermatologist and who require hospitalization will have their transition to the Emergency Department managed by the dermatologist with notification of the patient"s PCP. These patients who have follow-up in dermatology clinic will not require a follow-up visit with their primary care physician. The skin and lymph node exam performed by the dermatologist on patients in the treatment group will be documented in the electronic medical record for the subjects" medical records. Patients who are admitted after the initial outpatient discharge or at the follow-up visit will be considered treatment failures. A medical record review will be performed for patients in the treatment group two weeks after initial evaluation at the internal medicine clinic. A medical record review will be performed for patients who are randomized to the treatment group two weeks after initial evaluation at the internal medicine clinic.

Those in the control group who do not obtain a dermatology evaluation will follow primary care recommendations alone and will also have chart review two weeks later to assess for admission versus discharge home from clinic and outcome. In the control group, the need for additional clinical follow-up will be at the primary care physician"s discretion. These patients will receive a followup telephone call to confirm the final outcome of their condition two weeks after their visit to internal medicine clinic. The data sets generated from the treatment and control groups will then be compared to look for differences in hospital admission rates. For the treatment arm of the study, this data will be obtained during the follow-up visit and the medical record review. For the control arm, this will be obtained during both the medical record review and the follow-up phone call. The goal of this data collection is to determine what the final outcome is for patients in both groups in terms of need for hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign informed consent.
* Able to complete study and comply with study procedures.
* Presumed clinical diagnosis of cellulitis by primary care physician

Exclusion Criteria:

* Have a known postoperative site infection or abscess
* Have a human/animal bite
* Have known osteomyelitis
* Have a hardware/line infection
* Are under the age of 18
* Have a history of transplantation less than six months after initial transplant and/or if they have had an episode of acute rejection in the last 90 days
* Known use of antithymocyte globulin or campath in the last 6 months or more than 20 mg/day of prednisone for more than 30 days
* Are a known prisoner.
* Are decisionally-impaired.
* Have abnormal vital signs defined as systolic blood pressure <90 mmHg, diastolic blood pressure <80 mmHg, heart rate greater than 90 beats per minute or less than 50 beats per minute, respiratory rate greater than 20, or temperature > 100.5 F.
* Are known to be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of Hospital admission | 1 year

SECONDARY OUTCOMES:
Number of patients antibiotic was prescribed, type, dose, and duration of antibiotic prescribed and adverse events related to antibiotic usage. | 3 months
  We will be recording whether an antibiotic was prescribed, which antibiotic was used, the duration of treatment, the dosage of antibiotic, the cost of the antibiotic, and any adverse events related to antibiotic usage.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Kroshinsky, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Arakaki RY, Strazzula L, Woo E, Kroshinsky D. The impact of dermatology consultation on diagnostic accuracy and antibiotic use among patients with suspected cellulitis seen at outpatient internal medicine offices: a randomized clinical trial. JAMA Dermatol. 2014 Oct;150(10):1056-61. doi: 10.1001/jamadermatol.2014.1085. PMID 25143179